CLINICAL TRIAL: NCT07214883
Title: UCF MammoChat: An AI-Driven Platform for Personalized Breast Cancer Patient Support -Image Repository
Brief Title: UCF MammoChat: Image Repository
Status: Recruiting | Type: Observational
Sponsor: University of Central Florida (Other)
Collaborators: Florida Department of Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: STUDY00008263
Record Dates: First submitted 2025-10-08; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer; Breast Cancer Awareness; Breast Cancer Detection; Breast Cancer Survivors; Breast Cancer Female; Breast Cancer Diagnosis
Keywords: Breast Cancer; Artificial Intelligence; AI
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast Cancer Patients: Patients who have a been diagnosed with breast cancer
  Interventions: Other: No Interventions
- Controls: No breast cancer diagnosis
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: No Interventions — No intervention for participants.

SUMMARY:
This study aims to develop AI models to better read diagnostic mammograms for various populations and types of breast cancer, using the images that participants donate and their responses from study questionnaire to improve patient outcomes. This study also aims to provide mammography images to participants.

DETAILED DESCRIPTION:
Breast cancer patients often face overwhelming emotional and practical challenges, from feeling isolated to struggling to find the right information or resources during their treatment and recovery. These barriers can greatly impact both their quality of life and the effectiveness of their care. Among all US women, breast cancer is the second most common cancer and the second most common cause of cancer death. Recent guidelines recommend screening mammography in healthy women starting at 40 years old. The goal of screening mammography is to catch pre-cancerous lesions earlier so there is a high false positive error rate by design to not miss even remotely suspicious lesions on imaging. As evidenced by epidemiological studies, overdiagnosis in breast cancer is now a problem where up to 50% of screened women will have a false positive mammogram interpretation in their lifetime. The psychological impact of the false positivity manifest has significantly increased anxiety among patients that are needlessly recalled for false positive mammogram screening. Moreover, imprecise mammography interpretation may set off a complex cascade of potentially downstream surgical procedures (such as biopsy or mastectomy) for localized disease versus medical interventions such as radiation or chemotherapy for more advanced diseases.

The Health Insurance Portability and Accountability Act (HIPAA) gives patients the right to share their clinical data via informed consent for meaningful use such as research to improve health outcomes. One way of supporting breast cancer patients is by making their mammograms available to them. This allows patients to see and share their images. Some patients may be deterred from obtaining their images from their imaging centers due to cost and as they have no way to view DICOM images. Therefore, this study seeks to provide the mammography images to the participants.

While there are many open-source AI algorithms to improve precision in mammography interpretation, there are widely discrepant outcomes in breast cancer due to a complex and multifactorial disease etiology of different patient populations including social determinants of health. A recent retrospective study found that the integration of AI algorithms performed significantly better than the standard model for predicting breast cancer risk at 0 to 5 years 8. However, the bias in training data used to develop AI has long been recognized as limitations to its widespread application to marginalized populations as recently evidenced by a class action lawsuit against United Healthcare claiming its AI algorithms denied coverage and thus care to black and brown patients at scale 9,10. Moreover, the most cutting-edge algorithms in the current age of generative AI may often make random errors that can be disastrous in a clinical scenario. AI models are not omniscient as there is great variability in humans. AI models may need to be enhanced for different populations (such as different racial groups, ages ranges, or ethnicities) or for different types of breast cancer. Therefore, there is a stark need for accessible patient populations to demonstrate the applicability of robust AI to a diverse US population.

Therefore, using the images that the patients donate, the study aims to build AI models that can better read diagnostic mammograms.

ELIGIBILITY:
Inclusion Criteria:

* Adults, ages 18 and older
* Had a radiographic breast cancer imaging test, either for screening or diagnosis of breast cancer, with either positive or negative results performed in a US institution.
* Have an email account with access to a reliable internet connection or smartphone
* Pregnant women may choose to participate.

Exclusion Criteria:

* Minors , ages under 18
* Prisoners
* Adults who are unable to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be enrolled online from across the US. All study procedures are completed online. Potential participants will not be screened for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
AI model training using mammograms | 1 year
  Train, test and validate AI models with de-identified mammograms collected from imaging facilities.
Provide mammography images to participants | 1 year
  Once images are received, participant will have access to view their mammograms.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Gibson, PhD, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States